CLINICAL TRIAL: NCT04109677
Title: AIM CONTROL and the SWEdish CONcussion Study in Elite Handball (SWECON - Handball)
Brief Title: AIM CONTROL and SWECON - Handball The SWEdish CONcussion Study in Elite Handball
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Linkoeping University (Other Government)
Collaborators: Swedish Handball Federation (Unknown)
Responsible Party: Principal Investigator, Kajsa Johansson, Associate professor, senior lecturer, Linkoeping University
Other Study IDs: 88008-KJ-AIMCONTROL-SWECON
Record Dates: First submitted 2019-09-13; First posted 2019-09-30 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Sports Injuries; Concussion, Brain; Exposure; Psychological; Sports Physical Therapy
Keywords: Handball, sport injuries, concussion, acute overload injury
MeSH Terms: conditions — Athletic Injuries; Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SHE player: Female player in the top Swedish handball league
- Handbollsligan player: Male player in the top Swedish handball league

SUMMARY:
Handball is reported to be top 5 in Europe when it comes to sports injuries. There are few studies based on player reported data, and earlier Swedish data is mainly based on data from Insurance ´companies and mostly acute injuries. Earlier data lack the overuse injuries and number of injuries are taught to be underreported.

This epidemiological study has the objective to create research based knowledge about the injury panorama within Swedish handball with special interest in head-injuries in the elite level.

By using a mobile application "AIM Control", a retrospective weekly registration of handball related injuries was recorded together with self-assessed injury impact. Also data about sports/exercise exposure, other causes that could affect the players ability to practice/play matches, self-rated recovery before next practice/match as well as positive and negative affects will be analyzed.

Special emphasis is given to self-reported head injuries and the symptoms that the player might experience during the handball season 2019/2020. Data about symptom severity will be collected and analyzed together with AIM Controls other variables i.e. duration of symptoms and time to return-to-play. In case of a head-injury the Medical support team is contacted in order to describe the event, and interviewed with standardized questions about their thinking and action about how head injuries should be managed and prognosis of time to recovery and how to decide when a player is ready to play again? This is part of the AIM Control study called SWECON - handball.

DETAILED DESCRIPTION:
In co-operation with the Swedish Handball Federation, Swedish elite players are invited to participate during September 2019 and start to use the mobile application weekly during the current season (2019 to 2020.

By an electronic signed agreement, they receive unique user-name and log in. Download the free app from AppStore or Google Play, and then they are ready to start registration with questions in order to get retrospective data from the last week.

It takes 2-8 minutes to complete a registration, depending on if they have had a injury to report or not.

The data are stored according to data-regulations and GDPR on a secure server at Linköping University.

Players in the top League in Swedish handball, for the men called Handbollsligan and for females called SHE, together with contact persons for their Medical team will take part in the study. The later only when it comes to analysis of management of a head injury/concussion in case of such an injury in their team.

There is 14 possible male-teams within Handbollsligan and 12 possible female-team in SHE. Assessed possible number of players to register as a user of AIM Control is thought to be between 15-25 players peer team. Considering that some of them will not agree to participate or complete the study, a probable total number of participants might be 150 players in analysis.

This epidemiological study has the objective to create research based knowledge about the injury panorama within Swedish handball with special interest in head-injuries in the elite level.

A retrospective weekly registration by the handball player to record handball related injuries together with self-assessed injury impact. The application will push notice when it is time to do the weekly registration as well as a reminder.

Also data about sports/exercise exposure, other causes that could affect the players ability to practice/play matches, self-rated recovery before next practice/match as well as positive and negative affects will be analyzed.

If power, association between variables before injury occurs as well as afterwards is taught to be analyzed.

If a head injury is reported, possible symptoms afterwards will be self-reported in the app (part 2 in SCAT 5), and duration and when they return to team practice will be analyzed. Several questions regarding standard management and decisions for return to play is monitored by interviewing members of the Medical team and a follow-up interview with players with a handball related head-injury is planned to map retrospective experiences.

ELIGIBILITY:
Inclusion Criteria:

Player in the top league in Swedish handball (both men and women).

Exclusion Criteria:

* don´t read Swedish (the app:s language is Swedish)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Players in the top League in Swedish handball fort both men (called Handbollsligan) and women (called SHE) together with contact persons for the Medical team.
  There are 14 possible teams within Handbollsligan and 12 possible teams in SHE. The assessed possible number of players to register as a user of AIM Control is thought to be between 15-25 players per team. The total number of participants completing the study and possible for inclusion in the analysis is approximated to around 150 players.
  .
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Handball related injuries - prevalence/incidence | Weekly assessment during the handball season 2019 to 2020, retrospective related to the past week. Analyzed due to whole and part of the season.
  Self-rated injury/injuries in three categories:
  acute injury; earlier acute injury - still with symptoms; overload injury and their location.
  In relation to this, self-assessed impact in three perspectives (graded, ordinal scale):
  * participation in handball or handball related activities,
  * performance and
  * pain assessment. (Descriptive data, sub-categories.)
Focus: number of concussions (prevalence/incidence), severity of symptoms and duration, proportion due to other handball injuries, | Weekly assessment during the handball season 2019 to 2020, retrospective related to the past week. Analyzed due to whole and part of the season.
  Amount of concussions together with symptoms and duration. Using part of SCAT 5 - the "Symptom evaluation" together with analysis of return to play.
  Self-assessed impact of concussion in three perspectives (graded, ordinal scale):
  * participation within handball or handball related activities,
  * performance and
  * pain assessment. Descriptive data, sub-categories. Comparison with other injuries among handball players.

SECONDARY OUTCOMES:
12-item PANAS recording Positive and negative affects - relationship to injury or not | Weekly assessment during the handball season 2019 to 2020, retrospective related to the past week.
  Six positive and six negative affects (in each 3 activating and 3 deactivating) assessed weekly (range from a score 0-10). In case of injury analyze relationship before or after injury.
Exposure exercises/sports specific load due to practice sessions and matches and self assessed recovery - relationship to injury or not | Weekly assessment during the handball season 2019 to 2020, retrospective related to the past week
  Load in time for both handball related practice (in hours summeraized for the past week) and matches ( (in minutes of play summeraized for the past week) together with self-rated recovery before next handball session.
Injury analysis of a head trauma/concussion and related management within the handball teams medical support | The handball season 2019 to 2020 - performed consequently in teams with a player reported head injury.
  Answers and statements to a telephone questionnaire with medical team members. Open and closed answers about head injury situation within handball. Results in a case for questions about their reasoning about standard management, actions, both in the acute phase and during rehab. Decision making for return to play after head injury/concussion.

CONTACTS AND LOCATIONS:
Overall Officials: Kajsa Johansson, Ass.Prof., Principal Investigator — Linköping University, div. of Physiotherapy
Locations (1):
- Linköping University, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No